CLINICAL TRIAL: NCT01098162
Title: A Non-interventional Post-marketing Study, Evaluating Seizure Control and Tolerability of Vimpat® as Adjunctive Therapy to One Baseline Antiepileptic Drug in Epilepsy Patients With Partial-onset Seizures With or Without Secondary Generalization in Daily Clinical Practice in Germany
Brief Title: Vimpat® Added as Adjunctive Therapy to One Baseline Antiepileptic Drug
Acronym: VITOBA
Status: Completed | Type: Observational
Sponsor: UCB Pharma GmbH (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: SP0973
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Results first posted 2014-07-22 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Epilepsies, Partial
Keywords: Lacosamide; Vimpat®; Epilepsy; Partial-Onset Seizures; Adjunctive therapy
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vimpat®: Routine treatment in accordance with the local marketing authorization for Vimpat® added to one Baseline antiepileptic drug.

SUMMARY:
The purpose of this study is to systematically and prospectively collect data from patients with partial-onset seizures in routine clinical practice setting receiving adjunctive Vimpat®. The observed population will be only patients with one baseline antiepileptic drug. Seizure control and tolerability data will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The patient's treatment must be in accordance with the local marketing authorization (MA) for Vimpat®
* The decision to prescribe Vimpat® has to be made by the physician before and independently of his/her decision to include the patient in the study
* The Vimpat® treatment should have been started not longer than 2 weeks before study inclusion of the patient
* The patient must have a diagnosis of Epilepsy with Partial-Onset Seizures
* Based on the physician's clinical judgment, the patient's seizure activity is not controlled sufficiently on a current monotherapy and it is in the patient's best interest to be prescribed adjunctive Vimpat®

Exclusion Criteria:

In accordance with the Summary of Product Characteristics (SmPC)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Partial-Onset Seizures not sufficiently controlled with one Baseline Antiepileptic Drug (AED), treated by Epilepsy centers, clinics or office-based neurologists with adjunctive Vimpat® in routine daily practice.
Sampling Method: Non-Probability Sample
Enrollment: 576 (Actual)
Dates: Start 2010-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (113):
- Germany (113):
  - 55, Aachen
  - 119, Aalen
  - 194, Aichach
  - 191, Altenburg
  - 136, Alzenau in Unterfranken
  - 78, Aschaffenburg
  - 35, Bad Berka
  - 90, Baesweiler
  - 107, Berlin
  - 10A, Berlin
  - 141, Berlin
  - 25, Berlin
  - 49, Berlin
  - 66, Berlin
  - 75, Berlin
  - 36, Bielefeld
  - 5, Bonn
  - 192, Böblingen
  - 175, Brandenburg
  - 105, Chemnitz
  - 176, Cologne
  - 180, Cologne
  - 182, Coppenbrügge
  - 161, Dortmund
  - 128, Dresden
  - 21, Dresden
  - 39, Dresden
  - 111, Düren
  - 38, Düsseldorf
  - 7, Eberswalde
  - 102, Eisenach
  - 174, Eisenach
  - 56, Ellwangen
  - 50, Erbach im Odenwald
  - 179, Erfurt
  - 186, Erfurt
  - 6, Erlangen
  - 12, Essen
  - 27, Freiburg im Breisgau
  - 137, Fulda
  - 112, Gelsenkirchen
  - 103, Gera
  - 158, Göttingen
  - 65, Göttingen
  - 88, Göttingen
  - 1, Greifswald
  - 47, Grevenbroich
  - 134, Halle
  - 160, Hamburg
  - 71, Hamburg
  - 93, Hamm
  - 147, Heilbronn
  - 122, Herborn
  - 15, Herdecke
  - 130, Höchberg
  - 40, Immenstadt im Allgäu
  - 52, Jena
  - 61, Jülich
  - 44, Karlstadt am Main
  - 133, Kastellaun
  - 125, Kaufbeuren
  - 16, Kiel
  - 99, Kleve
  - 37, Krefeld
  - 46, Lappersdorf
  - 113, Leipzig
  - 4, Leipzig
  - 68, Leipzig
  - 81, Leipzig
  - 138, Lohr a. Main
  - 131, Ludwigsburg
  - 148, Lüdenscheid
  - 33, Mainz
  - 154, Mannheim
  - 151, Mühlhausen
  - 101, München
  - 167, München
  - 2, München
  - 43, Neuburg am Inn
  - 62, Neukirchen-Vluyn
  - 123, Neumarkt
  - 69, Nuremberg
  - 80, Oelde
  - 98, Oldenburg
  - 87, Oranienburg
  - 57, Potsdam
  - 3, Radeberg
  - 159, Rathenow
  - 45, Ravensburg
  - 95, Rostock
  - 85, Rüsselsheim am Main
  - 20, Schleswig
  - 157, Schlüchtern
  - 166, Schorndorf
  - 181, Schriesheim
  - 150, Schwäb. Gmünd
  - 168, Schwedt
  - 140, Senftenberg
  - 164, Siegen
  - 144, Sondershausen
  - 127, Stralsund
  - 14, Stuttgart
  - 170, Stuttgart
  - 104, Traunstein
  - 183, Troisdorf
  - 17, Tübingen
  - 13, Ulm
  - 48, Ulm
  - 54, Unterhaching
  - 171, Wermsdorf
  - 143, Westerstede
  - 79, Wismar
  - 169, Wolfratshausen

REFERENCES:
- [Derived] Runge U, Arnold S, Brandt C, Reinhardt F, Kuhn F, Isensee K, Ramirez F, Dedeken P, Lauterbach T, Noack-Rink M, Mayer T. A noninterventional study evaluating the effectiveness and safety of lacosamide added to monotherapy in patients with epilepsy with partial-onset seizures in daily clinical practice: The VITOBA study. Epilepsia. 2015 Dec;56(12):1921-30. doi: 10.1111/epi.13224. Epub 2015 Nov 3. PMID 26526971
- See also: Product Information — http://www.vimpat.com/pdf/PI.pdf
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This observational study started to enroll subjects in March 2010 in order to end up with 113 centers with enrolled subjects in Germany.
Pre-assignment Details: Participant Flow refers to the Enrolled Set (ES). The ES comprises all subjects who have been included in the observational study and for whom baseline examination data are available. Three patients were removed from the Enrolled Set after discussion in the Data Review Meeting.
Period: Overall Study
Arm/Group | Vimpat®
Started | 573
Completed | 461
Not Completed | 112
Not completed — Adverse Event | 37
Not completed — Lack of Efficacy | 4
Not completed — Wish of Patient | 7
Not completed — Lost to Follow-up | 9
Not completed — Lack of Efficacy & Wish of Patient | 5
Not completed — Adverse Event & Lack of Efficacy | 6
Not completed — Adverse Event & Wish of Patient | 13
Not completed — Adverse Event & Lost to Follow-up | 2
Not completed — AE & Lack of Efficacy & Wish of Patient | 1
Not completed — Wish of Patient & Lost to Follow-up | 1
Not completed — Other Reason | 1
Not completed — Reason Unknown | 26

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refer to the Full Analysis Set (FAS) which comprises all patients who have been treated with Vimpat® at least once and for whom a valid value of seizure frequency is available.
Arm/Group | Vimpat®
Number analyzed (Participants) | 520
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (17.0)
Age, Customized [Number; unit: participants]
  < 16 years | 0
  >= 16 years to <= 18 years | 7
  > 18 years to <= 64 years | 419
  >= 65 years | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 264
  Male | 256
Race/Ethnicity, Customized [Number; unit: participants]
  North/Middle European | 484
  South European | 28
  Asiatic | 3
  Arabic | 2
  Black African | 0
  Other Race | 3
Region of Enrollment [Number; unit: participants]
  Germany | 520

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression of Change (CGI-C) at Month 6
Description: For the assessment of the Clinical Global Impression of Change (CGI-C), the investigator provided his/her assessment of the subject's clinical status compared to Baseline. He/she was asked to check the category that best describes the subject's condition over the past 6 months compared to Baseline:
  * Very much improved
  * Much improved
  * Minimally improved
  * No change
  * Minimally worse
  * Much worse
  * Very much worse
Time Frame: Month 6
Population: Of the 520 subjects in the Full Analysis Set (FAS), 515 subjects are included in the analysis of this outcome measure.
  FAS comprises all subjects who have been treated with Vimpat® at least once, who fulfill the inclusion criteria and for whom a valid baseline and post-baseline value of seizure frequency is available.
Measure: Number; unit: participants
Arm/Group | Vimpat®
Number analyzed (Participants) | 515
participants
  Very Much Improved | 160
  Much Improved | 179
  Minimally Improved | 66
  No Change | 72
  Minimally Worse | 16
  Much Worse | 9
  Very Much Worse | 2
  Missing | 11

2. Secondary Outcome: Change in Number (Frequency) of Partial-onset Seizures Without Secondary Generalization From Baseline to Month 3
Description: Baseline values for the seizure frequency (SF) during the 12 weeks time period prior to inclusion ('historical baseline'), and the post-baseline values of seizure frequency reported after 3 months were normalized to a 28 days interval.
  Change in number of partial-onset seizures was derived as follows:
  Change in SF per 28 days = (SF at 3 months per 28 days) - (SF at Baseline per 28 days).
  A negative value in change from Baseline means that the value has decreased from Baseline to Month 3.
  Partial-onset seizures can be classified into one of the following three groups:
  * Simple partial seizures
  * Complex partial seizures
  * Partial seizures evolving to secondarily generalized seizures.
Time Frame: From Baseline to Month 3
Population: Of the 520 subjects in the Full Analysis Set (FAS), 449 subjects are included in the analysis of this outcome measure.
  FAS comprises all subjects who have been treated with Vimpat® at least once, who fulfill the inclusion criteria and for whom a valid baseline and post-baseline value of seizure frequency is available.
Measure: Mean (Standard Deviation); unit: Seizures per 28 days
Arm/Group | Vimpat®
Number analyzed (Participants) | 449
Seizures per 28 days | -3.80 (26.23)

3. Secondary Outcome: Change in Number (Frequency) of Partial-onset Seizures Without Secondary Generalization From Baseline to Month 6
Description: Baseline values for the seizure frequency (SF) during the 12 weeks time period prior to inclusion ('historical baseline'), and the post-baseline values of seizure frequency reported after 6 months were normalized to a 28 days interval.
  Change in number of partial-onset seizures was derived as follows:
  Change in SF per 28 days = (SF at 6 months per 28 days) - (SF at Baseline per 28 days).
  A negative value in change from Baseline means that the value has decreased from Baseline to Month 6.
  Partial-onset seizures can be classified into one of the following three groups:
  * Simple partial seizures
  * Complex partial seizures
  * Partial seizures evolving to secondarily generalized seizures.
Time Frame: From Baseline to Month 6
Population: Of the 520 subjects in the Full Analysis Set (FAS), 500 subjects are included in the analysis of this outcome measure.
  FAS comprises all subjects who have been treated with Vimpat® at least once, who fulfill the inclusion criteria and for whom a valid baseline and post-baseline value of seizure frequency is available.
Measure: Mean (Standard Deviation); unit: Seizures per 28 days
Arm/Group | Vimpat®
Number analyzed (Participants) | 500
Seizures per 28 days | -4.24 (26.22)

4. Secondary Outcome: Change in Number (Frequency) of Seizures With Secondary Generalization From Baseline to Month 3
Description: Baseline values for the seizure frequency (SF) during the 12 weeks time period prior to inclusion ('historical baseline'), and the post-baseline values of seizure frequency reported after 3 months were normalized to a 28 days interval.
  Change in number of partial-onset seizures with secondary generalization was derived as follows:
  Change in SF per 28 days = (SF at 3 months per 28 days) - (SF at Baseline per 28 days).
  A negative value in change from Baseline means that the value has decreased from Baseline to Month 3.
  Partial-onset seizures with secondary generalization can be classified into one of the following three groups:
  * Simple partial seizures evolving to generalized seizures
  * Complex partial seizures evolving to generalized seizures
  * Simple partial seizures evolving to Complex partial seizures evolving to generalized seizures.
Time Frame: From Baseline to Month 3
Population: Of the 520 subjects in the Full Analysis Set (FAS), 447 subjects are included in the analysis of this outcome measure.
  FAS comprises all subjects who have been treated with Vimpat® at least once, who fulfill the inclusion criteria and for whom a valid baseline and post-baseline value of seizure frequency is available.
Measure: Mean (Standard Deviation); unit: Seizures per 28 days
Arm/Group | Vimpat®
Number analyzed (Participants) | 447
Seizures per 28 days | -0.39 (1.61)

5. Secondary Outcome: Change in Number (Frequency) of Seizures With Secondary Generalization From Baseline to Month 6
Description: Baseline values for the seizure frequency (SF) during the 12 weeks time period prior to inclusion ('historical baseline'), and the post-baseline values of seizure frequency reported after 6 months were normalized to a 28 days interval.
  Change in number of partial-onset seizures with secondary generalization was derived as follows:
  Change in SF per 28 days = (SF at 6 months per 28 days) - (SF at Baseline per 28 days).
  A negative value in change from Baseline means that the value has decreased from Baseline to Month 6.
  Partial-onset seizures with secondary generalization can be classified into one of the following three groups:
  * Simple partial seizures evolving to generalized seizures
  * Complex partial seizures evolving to generalized seizures
  * Simple partial seizures evolving to Complex partial seizures evolving to generalized seizures.
Time Frame: From Baseline to Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Seizures per 28 days
Arm/Group | Vimpat®
Number analyzed (Participants) | 500
Seizures per 28 days | -0.39 (1.88)

6. Secondary Outcome: Incidence of Adverse Events During the Study
Description: The number of subjects affected by any Treatment Emergent Adverse Event (TEAE) during the course of the study from Day 0 up to Month 6 is presented below.
Time Frame: From Inclusion Visit (Day 0) up to Month 6
Population: All 571 subjects in the Safety Set are included in the analysis of this outcome measure.
  Safety Set comprises all patients included who have been treated with Vimpat® at least once.
Measure: Number; unit: participants
Arm/Group | Vimpat®
Number analyzed (Participants) | 571
participants | 277

ADVERSE EVENTS:
Time Frame: Adverse Events were collected during the whole study from Inclusion Visit (Day 0) up to Month 6.
Description: Adverse Events refer to the Safety Set, which comprises all enrolled subjects who have been treated with Vimpat at least once.
Arm/Group | Vimpat®
Serious Adverse Events (participants affected / at risk) | 56/571
Other Adverse Events (participants affected / at risk) | 114/571
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vimpat® (N=571)
Angina pectoris (Cardiac disorders) | 2 (3)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Renal function test abnormal (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Convulsion (Nervous system disorders) | 10 (11)
Grand mal convulsion (Nervous system disorders) | 9 (10)
Epilepsy (Nervous system disorders) | 7 (9)
Dizziness (Nervous system disorders) | 5 (5)
Status epilepticus (Nervous system disorders) | 4 (5)
Syncope (Nervous system disorders) | 4 (4)
Brain stem ischaemia (Nervous system disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Nystagmus (Nervous system disorders) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1)
Postictal paralysis (Nervous system disorders) | 1 (1)
Postictal state (Nervous system disorders) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Conversion disorder (Psychiatric disorders) | 3 (3)
Disorientation (Psychiatric disorders) | 2 (2)
Acute psychosis (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 1 (1)
Mood swings (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Acute prerenal failure (Renal and urinary disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vimpat® (N=571)
Fatigue (General disorders) | 71 (75)
Dizziness (Nervous system disorders) | 60 (69)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days